CLINICAL TRIAL: NCT05793437
Title: Effects of Permissive Hypercapnia on Concentration of Postoperative Plasma Neurofilament Light in Elderly Patients Undergoing Laparoscopic Surgery:A Prospective, Randomized Controlled Study
Brief Title: Effects of Permissive Hypercapnia on Concentration of Postoperative Plasma Neurofilament Light
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Principal Investigator, Qing-he Zhou, Principal investigator, Affiliated Hospital of Jiaxing University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-KY-050
Record Dates: First submitted 2023-03-03; First posted 2023-03-31 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Hypercapnia
Keywords: Neurofilament light; Hypercapnia
MeSH Terms: conditions — Hypercapnia; Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- permissive hypercapnia (Experimental): Tidal volume (6-8ml/kg) and respiratory rate is adjusted to achieve the objective values of PaCO2:45～55mmHg
  Interventions: Behavioral: permissive hypercapnia
- normocapnia (Active Comparator): Tidal volume (8-10ml/kg) and respiratory rate is adjusted to achieve the objective values of PaCO2:35～45mmHg
  Interventions: Behavioral: normocapnia

INTERVENTIONS:
Behavioral: permissive hypercapnia — Tidal volume (6-8ml/kg) and respiratory rate is adjusted to achieve the objective values of PaCO2:45～55mmHg
  Other Names: PaCO2:45～55mmHg
  Arms: permissive hypercapnia
Behavioral: normocapnia — Tidal volume (8-10ml/kg) and respiratory rate is adjusted to achieve the objective values of PaCO2:35～45mmHg
  Other Names: PaCO2:35～45mmHg
  Arms: normocapnia

SUMMARY:
The aim of this study is to conduct a prospective, single-center randomized controlled study to investigate the changes of plasma NFL concentration in patients undergoing laparoscopic surgery with mild hypercapnia, and further explore its impact on the central nervous system.

DETAILED DESCRIPTION:
Plasma NFL concentrations were measured preoperatively and 1 day postoperatively.

Secondary endpoints:CAM (Confusion Assessment Method) is conducted to check the subjects' baseline cognitive function preoperative day and 1 day postoperatively to assess whether delirium occurs.

ELIGIBILITY:
Inclusion Criteria:

* age over 60 years
* duration of pneumoperitoneum greater than 60 minutes
* American Society of Anesthesiology (ASA) status Ⅱ-Ⅲ
* undergoing laparoscopic surgery under general anesthesia with endotracheal intubation

Exclusion Criteria:

* history of mental or neurological disorders
* preoperative use of antipsychotic drugs
* American Society of Anesthesiology (ASA) status Ⅳ
* severe abnormalities in heart, lung, liver, kidney, and coagulation function
* Intracranial space-occupying lesions or major cerebrovascular diseases (such as carotid atherosclerosis and cerebral aneurysm)
* Severe hypertension or hypotension
* Severe metabolic acidosis or hypercapnic respiratory failure before surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-01-28 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
Changes in plasma Neurofilament Light levels | 1 week
  Comparison of changes in plasma Neurofilament Light levels pre and postoperative in patients exposed and not exposed to hypercapnia.

CONTACTS AND LOCATIONS:
Overall Officials: Qinghe Zhou, Principal Investigator — Affiliated Hospital of Jiaxing University
Locations (1):
- Affiliated Hospital of Jiaxing University, Jiaxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No